CLINICAL TRIAL: NCT00576017
Title: Randomised Study to Evaluate the Efficacy and Safety of Fentanyl-TTS Versus Weak Opioids in Patients With Moderate to Severe Chronic Cancer Pain Previously Treated With NSAIDs (Non-steroidal Anti-inflammatory Drugs).
Brief Title: A Study to Evaluate the Safety and Effectiveness of Fentanyl-TTS Compared to Weak Opioids in Patients With Moderate to Severe Chronic Cancer Pain Previously Treated With NSAIDS (Non-steroidal Anti-inflammatory Drugs).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag, S.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003526
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Pain
Keywords: Cancer pain treatment; Fentanyl TTS; Dihydrocodeine; Tramadol; Cancer pain; Durogesic; Ultram
MeSH Terms: conditions — Pain; Cancer Pain

INTERVENTIONS:
Drug: Fentanyl-TTS

SUMMARY:
To show, using the analgesic WHO scale, that fentanyl-TTS may be directly used for treating moderate to severe cancer pain in patients treated with NSAIDs, acetaminophen, or metamizole (first step drugs) avoiding the second step, and may be at least as effective and safe as currently used second step drugs, minor opioids.

DETAILED DESCRIPTION:
This study is a multicenter, randomized(study drug assigned by chance), open-label, nationwide study. Patients with moderate to severe chronic pain due to the oncological disease (VAS>5) meeting the inclusion and exclusion criteria were randomized to treatment with fentanyl-TTS (transdermal patches, initial dosage: 25µg/h patch every 3 days, experimental drug) or with minor opioids (Tramadol, initial dosage of 200mg/day and Dihydrocodeine initial dosage of 120mg/day, control arm). The follow-up and drug administration was two months, during which controls were performed every 7 days, except for the first that was on Day 4. If pain was not controlled (VAS<3), the investigator could increase the dose of the relevant drug (according to data sheet). The primary endpoint has been the control of pain during treatment. Pain was assessed by the visual analogue scale. Pain severity was assessed at each follow-up visit. The secondary endpoint was to assess the advantages of using fentanyl-TTS after the first step of the WHO analgesic ladder as compared to minor opioids. These advantages were assessed based on the incidence of side effects associated with treatment with opioids during treatment where the following was assessed by a table with the most common side effects: nausea, vomiting, constipation and drowsiness (WHO) and their severity, the quantity of support drugs required by the patients to cope with the side effects occurring, adverse events related to the study drug, and the percentage of patients discontinuing or switching treatment due to side effects. Fentanyl, dosage forms: 25µg/h, 50µg/h and 100µg/h. Transdermal patches (initial dosage: 25µg/h patch every 3 days). Tramadol, dosage forms: 100mg, 150mg and 200mg, (initial dosage: 200mg/day). Dihydrocodeine, dosage forms: 60mg, 90mg and 120mg, (initial dosage: 120mg/day). If pain was not controlled (VAS<3), the investigator could increase the dose of the relevant drug. The follow-up and drug administration was two months, during which controls were performed every 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe chronic pain due to the oncological condition, defined as VAS => 5, treated with first step drugs, either NSAIDs or acetaminophen or metamizole (the dose of first step drugs requiring a switch in treatment is left to the physician's discretion)
* Patients with a documented histological diagnosis of cancer.

Exclusion Criteria:

* Patients whose pain has some neuropathic component
* Patients who have been treated with opioids during the 2 months prior to study entry
* Patients with dermatological disease, a history of allergy or hypersensitivity to fentanyl or to adhesive components preventing use of patches
* Patients with a history of cardiac, CNS, or respiratory disease that prevents their participation in the study in the investigator's judgment
* Patients with kidney or liver failure contraindicating use of opioids based on medical criterion
* Pregnant women or women of childbearing age who do not use an effective contraceptive method throughout the study
* Patients in whom surgery is planned during the study
* Patients who are participating at the same time in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-10; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the control of pain during treatment. Pain was assessed by the visual analogue scale. Pain severity was assessed at each follow-up visit.

SECONDARY OUTCOMES:
The secondary endpoint was to assess the advantages of using fentanyl-TTS after the first step of the WHO analgesic ladder as compared to minor opioids.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- See also: A study to evaluate the safety and effectiveness of fentanyl-TTS compared to weak opiods in patients with moderate to severe chronic cancer pain previously treated with NSAIDS (non-steroidal anti-inflammatory drugs). — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=278&filename=CR003526_CSR.pdf